CLINICAL TRIAL: NCT02978092
Title: Monochromatic Digital-Pupillometry With Two Automated Devices in Comparison to Manual Measurements on Digital Photographs
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Dr. Martin Leitritz, PD Dr. med., University Hospital Tuebingen
Other Study IDs: 3
Record Dates: First submitted 2016-11-26; First posted 2016-11-30 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Pupil Examination

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Retrospective, analysis of three different methods to measure patients' pupil diameters

ELIGIBILITY:
Inclusion Criteria:

* usable measurement values from three different examinations

Exclusion Criteria:

* bad image quality

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients of a university eye-hospital which underwent examinations for refractive or cataract surgery
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2016-04; Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Pupils' diameter | September 2016
  Measurement of patients pupil diameter with several methods